CLINICAL TRIAL: NCT04846647
Title: Study of the Inappropriate Secretion of FGF23 in Patients Followed in Hospital in a Context of Hypophosphatemia
Acronym: IFEH
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: DiaSorin ; Saluggia, Italia (Unknown)
Responsible Party: Sponsor
Other Study IDs: RNI 2021 BOUVIER; 2021-A00284-37 (Other: 2021-A00284-37)
Record Dates: First submitted 2021-04-13; First posted 2021-04-15 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Hypophosphatemia Without Immediate Anteriority; Unexplained Hypophosphatemia
Keywords: FGF-23; Unexplained hypophosphatemia; Phosphate metabolism; Physiopathology of hypophosphatemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Unexplained hypophosphatemia: Collection of additional blood volume (approximately 10 mL) during blood tests provided as part of the usual medical care.
  Interventions: Behavioral: unexplained hypophoshatemia

INTERVENTIONS:
Behavioral: unexplained hypophoshatemia — Collection of additional blood volume (approximately 10 mL) during blood tests provided as part of the usual medical care.

SUMMARY:
The discovery of FGF23, the missing link in the long researched and finally found phosphate metabolism, marked a turning point in the understanding and physiopathology of specific hypophosphatemia. By inhibiting the renal reabsorption of phosphate and the production of calcitriol, FGF23 behaves like a hypophosphatemia hormone.

Hypersecretion of FGF23 can occur in the case of genetic abnormalities (X-linked hypophosphatemic vitamin-resistant rickets, recessive or dominant hypophosphatemic rickets, McCune-Albright syndrome ...) or acquired abnormalities (oncogenic osteomalacia). Oncogenic osteomalacia can be induced by hyperproduction of FGF23 by benign tumours of mesenchymal origin. But more recently, several cases of malignant tumours secreting FGF23 have also been described (prostate, colon, breast, ovarian and lung cancers, pulmonary carcinoma, etc.)

DETAILED DESCRIPTION:
To date, even if the incidence of FGF23-secreting tumours seems rare, no precise bibliographical data is available in the scientific literature. Future studies will have to address this issue in order not to underestimate the frequency of this complication.

In this context, investigators would like to study the incidence of inappropriate FGF23 increase from a collection of biological samples carried out on 500 patients treated at the Clermont-Ferrand University Hospital for hypophosphatemia.

ELIGIBILITY:
Inclusion Criteria:

* Major patient, male or female
* Taken care of at the Clermont-Ferrand University Hospital or the Jean Perrin Centre
* In a context of hypophosphatemia (< 0.80 mmol/L), without immediate anteriority and not occurring during hospitalisation
* In capacity to express informed consent to participate in research
* Affiliated to a social security system

Exclusion Criteria:

* Previously diagnosed hypophosphatemia
* Hypophosphatemia during hospitalisation
* Haemodialysis patient
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Major patient, male or female with hypophosphatemia (< 0.80 mmol/L), without immediate anteriority
Sampling Method: Non-Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2021-10-05 (Actual); Primary Completion 2022-04-25 (Actual); Study Completion 2022-04-25 (Actual)

PRIMARY OUTCOMES:
Evaluate the frequency of blood levels of FGF23 unsuitable for hypophosphatemia | day 0
  Assessing the presence of a blood level of FGF23 considered unsuitable for hypophosphatemia

SECONDARY OUTCOMES:
Investigate the relationship between blood levels of FGF23 and other biochemical parameters in hospital patients with hypophosphatemia.. | Day 1
  Description: Measure blood levels of FGF23 in absolute value and other biochemical parameters (phosphatemia, phosphaturia, PTH, vitamin D ...)
Investigate the relationship between blood levels of FGF23 and other biochemical parameters in hospital patients with hypophosphatemia. | day 1
  Measure blood levels of FGF23 in absolute value and other biochemical parameters (phosphatemia, phosphaturia, PTH, vitamin D ...).

CONTACTS AND LOCATIONS:
Overall Officials: Damien BOUVIER, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (2):
- France (2):
  - Chu Clermont Ferrand, Clermont-Ferrand
  - Centre Jean Perrin, Clermont-Ferrand

REFERENCES:
- [Background] Suvannasankha A, Tompkins DR, Edwards DF, Petyaykina KV, Crean CD, Fournier PG, Parker JM, Sandusky GE, Ichikawa S, Imel EA, Chirgwin JM. FGF23 is elevated in multiple myeloma and increases heparanase expression by tumor cells. Oncotarget. 2015 Aug 14;6(23):19647-60. doi: 10.18632/oncotarget.3794. PMID 25944690
- [Background] Imel EA, Biggin A, Schindeler A, Munns CF. FGF23, Hypophosphatemia, and Emerging Treatments. JBMR Plus. 2019 May 13;3(8):e10190. doi: 10.1002/jbm4.10190. eCollection 2019 Aug. PMID 31485552
- [Background] Endo I, Fukumoto S, Ozono K, Namba N, Inoue D, Okazaki R, Yamauchi M, Sugimoto T, Minagawa M, Michigami T, Nagai M, Matsumoto T. Nationwide survey of fibroblast growth factor 23 (FGF23)-related hypophosphatemic diseases in Japan: prevalence, biochemical data and treatment. Endocr J. 2015;62(9):811-6. doi: 10.1507/endocrj.EJ15-0275. Epub 2015 Jul 1. PMID 26135520